CLINICAL TRIAL: NCT00113815
Title: A Randomized, Double-Blind, Placebo-Controlled, Fixed Dose-Ranging Study to Assess the Safety, Tolerability, and Efficacy of Topiramate Oral Liquid and Sprinkle Formulations as an Adjunct to Concurrent Anticonvulsant Therapy for Infants (1-24 Months of Age) With Refractory Partial-Onset Seizures
Brief Title: Topiramate as Adjunctive Therapy in Infants 1-24 Months for the Control of Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR002233
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Partial Seizure Disorder; Epilepsy; Seizures
Keywords: Partial seizure disorder; Topiramate; Epilepsy; Infants
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 003 (Experimental): topiramate 25 mg/kg/day
  Interventions: Drug: topiramate
- 002 (Experimental): topiramate 15 mg/kg/day
  Interventions: Drug: topiramate
- 001 (Experimental): topiramate 5 mg/kg/day
  Interventions: Drug: topiramate
- 004 (Experimental): placebo placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: topiramate — 15 mg/kg/day
  Arms: 002
Drug: topiramate — 5 mg/kg/day
  Arms: 001
Drug: topiramate — 25 mg/kg/day
  Arms: 003
Drug: placebo — placebo
  Arms: 004

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety and efficacy of topiramate in infants with refractory partial onset seizures (POS).

DETAILED DESCRIPTION:
This is a world wide, multicenter, randomized, double-blind, placebo-controlled study to evaluate the tolerability, safety and efficacy of 3 target doses (5, 15, and 25 mg/kg/day) of topiramate compared with placebo as an adjunct therapy in infants with refractory partial onset seizures (POS). There are 4 phases to the study, a screening phase of 3 days, a double blind treatment phase of 20 days, a one year open label extension phase and a posttreatment (taper and withdrawal) phase. The oral liquid formulation will also be assessed during this study, as it is investigational, unlike the marketed sprinkle formulation. 5, 15, 25 mg/kg/day of topriramate sprinkle and oral liquid formulation will be administered during the four phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1-24 months, inclusive
* Concurrent 1 or 2 antiepileptic drugs
* Receiving regular enteral feedings
* Weigh between 3.5 and 15 kg
* Clinical or EEG evidence of simple or complex POS

Exclusion Criteria:

* Exclusively breast fed and cannot take medicine by mouth
* Surgically implanted and functioning vagus nerve stimulator
* Renal stones
* Medically uncontrolled illnesses or conditions
* Infantile seizures as a result of a correctable medical condition
* Progressive neurologic disorder

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Video-recorded EEG was primary efficacy measure. Baseline vEEG and the vEEG at Visit 4 (Days 19 to 20; end point DB treatment phase or early withdrawal) will be read by a blinded central reader | Video-recorded EEG was primary efficacy measure. Baseline vEEG and the vEEG at Visit 4 (Days 19 to 20; end point DB treatment phase or early withdrawal) will be read by a blinded central reader

SECONDARY OUTCOMES:
Percent treatment responders >=50% reduction seizure rate. ·Percentage change in seizure rate recorded on subject take-home records. Percentage change in seizure rates for all seizure types recorded on VEEG. | Baseline to endpoint of double blind phase

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (94):
- United States (47):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Los Angeles, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Loxahatchee Groves, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Dearborn, Michigan
  - Saint Paul, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Cherry Hill, New Jersey
  - Newark, New Jersey
  - Buffalo, New York
  - Mineola, New York
  - Rochester, New York
  - Stony Brook, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Danville, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Fort Worth, Texas
  - Plano, Texas
  - Norfolk, Virginia
  - Madison, Wisconsin
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Rio Negro
  - Santa Fe
- Australia (3):
  - Heidelberg West
  - Melbourne
  - Subiaco
- Belgium (4):
  - Antwerp
  - Ghent
  - Leuven
  - Pulderbos
- Canada (2):
  - St. John's, Newfoundland and Labrador
  - Saskatoon, Saskatchewan
- Chile (2):
  - Chile
  - Santiago
- Finland (2):
  - Helsinki
  - Tampere
- France (3):
  - Bordeaux
  - Lille
  - Tours
- Budapest, Hungary
- India (6):
  - Chennai
  - Hyderabad Gpo
  - Kochi Ho
  - Mumbai
  - New Delhi
  - Pune
- Petah Tikva, Israel
- Mexico (2):
  - Monterrey
  - San Luis Potosí City
- Heeze, Netherlands
- Wellington, New Zealand
- Bergen, Norway
- Poland (2):
  - Gdansk
  - Warsaw
- Russia (4):
  - Ekaterinburg Siberia
  - Moscow
  - Omsk Siberia
  - Samara
- Cape Town Wc, South Africa
- Seoul, South Korea
- Madrid, Spain
- Taipei, Taiwan
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Ukraine (2):
  - Donetsk
  - Kiev

REFERENCES:
- [Result] Novotny E, Renfroe B, Yardi N, Nordli D, Ness S, Wang S, Weber T, Kurland CL, Yuen E, Eerdekens M, Venkatraman L, Nye JS, Ford L. Randomized trial of adjunctive topiramate therapy in infants with refractory partial seizures. Neurology. 2010 Mar 2;74(9):714-20. doi: 10.1212/WNL.0b013e3181d1cd4c. Epub 2010 Jan 20. PMID 20089937
- [Derived] Ness S, Todd MJ, Wang S, Eerdekens M, Nye JS, Ford L. Adaptive behavior outcomes in infants treated with adjunctive topiramate. Pediatr Neurol. 2012 Jun;46(6):350-8. doi: 10.1016/j.pediatrneurol.2012.02.028. PMID 22633629
- [Derived] Puri V, Ness S, Sattaluri SJ, Wang S, Todd M, Yuen E, Eerdekens M, Nye JS, Manitpisitkul P, Shalayda K, Ford L. Long-term open-label study of adjunctive topiramate in infants with refractory partial-onset seizures. J Child Neurol. 2011 Oct;26(10):1271-83. doi: 10.1177/0883073811406982. Epub 2011 Jun 14. PMID 21673279
- See also: Topiramate as Adjunctive Therapy in Infants 1-24 Months for the Control of Partial Onset Seizures — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=460&filename=CR002233_CSR.pdf